CLINICAL TRIAL: NCT02866383
Title: A Prospective Randomized, Open-label Phase 2 Study of Immune Checkpoint Inhibition, Nivolumab With or Without Ipilimumab in Combination With Radiation Therapy in Pretreated Patients With Metastatic Pancreatic Cancer or Biliary Tract Cancer.
Brief Title: Immune Checkpoint Inhibition in Combination With Radiation Therapy in Pancreatic Cancer or Biliary Tract Cancer Patients
Acronym: CheckPAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Inna Chen, MD, Staff Specialist, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GI 1616
Record Dates: First submitted 2016-08-08; First posted 2016-08-15 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Pancreatic Cancer; Metastatic Biliary Tract Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms | interventions — Nivolumab; Ipilimumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nivolumab & Radiotherapy (Experimental): Patients will receive nivolumab 3 mg/kg over 60 minutes as an IV infusion on day 1 just after RT and then every 2 weeks (q2w), for a maximum of 52 weeks
  Interventions: Drug: Nivolumab; Radiation: Radiotherapy
- Nivolumab & Ipilimumab & Radiotherapy (Experimental): Patients will receive nivolumab 3 mg/kg over 60 minutes as an IV infusion on day 1 just after RT. Thirty minutes after the completion of nivolumab infusion patients will receive ipilimumab 1 mg/kg over 90 minutes IV as an IV infusion. Nivolumab will be given every 2 weeks (q2w) and ipilimumab every 6 weeks (q6w), respectively for a maximum of 52 weeks
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Nivolumab — 3 mg/kg is given over 60 minutes I.V. on day 1 just after radiation and then every 2 weeks (q2w)
  Other Names: Opdivo®
Drug: Ipilimumab — 1 mg/kg is given over 90 minutes I.V. on day 1 30 minutes after the completion of nivolumab infusion and then every 6 weeks IV (q6w)
  Other Names: Yervoy®
  Arms: Nivolumab & Ipilimumab & Radiotherapy
Radiation: Radiotherapy — 15 Gy x 1 fraction given on day 1

SUMMARY:
This is a prospective, randomized, open-label phase 2 study in patients with metastatic PC or BTC refractory or intolerant to at least one line of prior systemic chemotherapy with gemcitabine or platinum-containing regimens to determine the efficacy and safety of nivolumab or nivolumab plus ipilimumab administered concurrently with high dose RT. Patients with metastatic PC or BTC who are feasible candidates for radiation and biopsy of primary and/or metastatic lesions will be included.

DETAILED DESCRIPTION:
This was a randomized phase II trial conducted at Herlev & Gentofte Hospital. Patients were stratified according to PS and randomized into two arms (1:1) (Appendix Figure A1 and Data Supplement, online only). Patients received SBRT consisting of 15 Gy (day 1) to a single primary or metastatic lesion with 3 mg/kg of intravenous nivolumab (IV) on day 1 and every 2 weeks (q2w) (Arm A), or SBRT consisting of 15 Gy (day 1) with 3 mg/kg of IV nivolumab (day 1) q2w and 1 mg/kg of IV ipilimumab on day 1 and every 6 weeks (Arm B).

A safety phase involving a run-in assessment of three patients from each arm (n = 6) was followed by the expansion phase. The patients were monitored for dose-limiting toxicities prior to the expansion. Treatment was continued for a maximum of 52 weeks or until progressive disease (PD), unacceptable toxicity, withdrawal of consent, or clear clinical deterioration according to the investigator's judgment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent

  * Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care
  * Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
* Histopathological confirmation of pancreatic adenocarcinoma or BTC prior to entering this study OR histopathological confirmation of carcinoma in the setting of clinical and radiological characteristics which, together with the pathology, are consistent with a diagnosis of PC or BTC
* At least one measurable primary in-situ (or locally-recurrent) or metastatic tumor must be present and, in the opinion of radiation oncologist, be amenable to RT as planned in the protocol and at least one additional metastatic tumor that will not undergo RT and which is measurable according to RECIST 1.1 criteria. Both lesions must be accessible for image-guided percutaneous biopsy
* There is no upper limit on the number of prior chemotherapy regimens received. Patients must have received and failed or intolerance to at least one line of prior systemic chemotherapy with gemcitabine or platinum-containing regimens for unresectable and/or metastatic PC or BTC
* Age > 18 years and older
* Life expectancy greater than 3 months
* ECOG/WHO Performance Status (PS) 0-1
* Patients must have normal organ and marrow function as defined below:
* White blood cell count (WBC) ≥ 2 x 10⁹/L
* Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L
* Hemoglobin ≥ 5,6 mmol/l
* Platelet count ≥ 100 x 10⁹/L
* Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) (patients with Gilbert's Syndrome must have a total bilirubin < 3.0 mg/dL)
* ASAT/ALAT ≤ 3 x ULN ( < 5 x ULN if known liver metastasis)
* PP ≥ 40 or INR ≤ 1.5
* Serum creatinine ≤ 1.5 x ULN or CrCl ≥ 40 mL/min (using the Cockcroft-Gault formula)
* Women of childbearing potential (WOCBP) must use method(s) of contraception as indicated per protocol. For a teratogenic study drug and/or when there is insufficient information to assess teratogenicity (preclinical studies have not been done), a highly effective method(s) of contraception (failure rate of less than 1% per year) is required. The individual methods of contraception and duration should be determined in consultation with the investigator. WOCBP must follow instructions for birth control when the half-life of the investigational drug is greater than 24 hours, contraception should be continued for a period of 30 days plus the time required for the investigational drug to undergo five half-lives. The half-life of nivolumab and ipilimumab is up to 25 days and 18 days, respectively. WOCBP should therefore use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug.
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab
* Women must not be breastfeeding
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year The investigator shall review contraception methods and the time period that contraception must be followed. Men that are sexually active with WOCBP must follow instructions for birth control when the half-life of the investigational drug is greater than 24 hours, contraception should be continued for a period of 90 days plus the time required for the investigational drug to undergo five half-lives. The half-life of nivolumab and ipilimumab is up to 25 days and 18 days, respectively. Men who are sexually active with WOCBP must continue contraception for 31 weeks (90 days plus the time required for nivolumab to undergo five half lives) after the last dose of investigational drug. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception
* Subjects must have signed and dated a BIOPAC IRB/IEC approved written informed consent form and patients with BTC must have signed and dated a CHOCA in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care

Exclusion Criteria:

* Malignant ascites that is clinically detectable by physical examination or is symptomatic. Evidence of radiographic ascites that is not clinically significant will not be exclusion criteria
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* No chemotherapy, radiotherapy, or major surgery within the last 2 weeks prior to entering the study
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results
* Patients should be excluded if they have an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Patients should be excluded if they are positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* As there is potential for hepatic toxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatoxicity should be used with caution in patients treated with nivolumab- and ipilimumab containing regimen
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Allergies and Adverse Drug Reaction

  * History of allergy to study drug components
  * History of severe hypersensitivity reaction to any monoclonal antibody
* WOCBP who are pregnant or breastfeeding
* Women with a positive pregnancy test at enrollment or prior to administration of study medication
* Patients are excluded if they have active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for [lowest minimum is 4 weeks or more] after treatment is complete and within 28 days prior to the first dose of nivolumab administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate (CBR) | 6 months
  Stable disease (SD) or complete response (CR) or partial response (PR)according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | 12 months
  Assessment based on AEs, SAEs, laboratory abnormalities
CBR | 6 months
  CBR according to modified immune-related Response Criteria (irRC)
Overall response rate (ORR) according to RECIST 1.1 | 6 months
  PR or CR according to RECIST 1.1
Overall response rate (ORR) according to modified irRC | 6 months
  PR or CR according to modified irRC
Progression free survival (PFS) per RECIST 1.1 | 6 months
  Time from the date of randomization until the date of PD determined by investigator assessment of objective radiographic disease assessments per RECIST 1.1, or death due to any cause if sooner
Progression free survival (PFS) per modified irRC | 6 months
  Time from the date of randomization until the date of PD determined by investigator assessment of objective radiographic disease assessments per modified irRC, or death due to any cause if sooner
Overall survival (OS) probability at 6 months | 6 months
  The Kaplan-Meier estimate of proportion of patients that survived from the date of randomization by 6 months
OS | 12 months
  Time from the date of randomization until death due to any cause
QoL | 12 months
  Quality of Life Questionnaire C30 Version 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Inna Chen, MD, Principal Investigator — Herlev and Gentofte Hospital
Locations (1):
- Herlev & Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johansen AZ, Novitski SI, Hjaltelin JX, Theile S, Boisen MK, Brunak S, Madsen DH, Nielsen DL, Chen IM. Plasma YKL-40 is associated with prognosis in patients with metastatic pancreatic cancer receiving immune checkpoint inhibitors in combination with radiotherapy. Front Immunol. 2023 Sep 7;14:1228907. doi: 10.3389/fimmu.2023.1228907. eCollection 2023. PMID 37744345
- [Derived] Chen IM, Johansen JS, Theile S, Hjaltelin JX, Novitski SI, Brunak S, Hasselby JP, Willemoe GL, Lorentzen T, Madsen K, Jensen BV, Wilken EE, Geertsen P, Behrens C, Nolsoe C, Hermann KL, Svane IM, Nielsen D. Randomized Phase II Study of Nivolumab With or Without Ipilimumab Combined With Stereotactic Body Radiotherapy for Refractory Metastatic Pancreatic Cancer (CheckPAC). J Clin Oncol. 2022 Sep 20;40(27):3180-3189. doi: 10.1200/JCO.21.02511. Epub 2022 Apr 27. PMID 35476508